CLINICAL TRIAL: NCT01587586
Title: An Open-label, Randomized, Active Control Study to Evaluate the Antiviral Activity, Safety and Pharmacokinetics of P1101 + Ribavirin in Treatment-Naïve Subjects With HCV Genotype 1 Infection
Brief Title: Dose Finding Study of Pegylated-P-Interferon-alpha-2b(P1101) in Treatment-Naive Subjects With Hepatitis C Virus Genotype 1 Infection
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: PharmaEssentia (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A11-201
Record Dates: First submitted 2012-04-26; First posted 2012-04-30 (Estimated); Last update posted 2021-10-15 (Actual); Status verified 2021-10

CONDITIONS: Hepatitis C, Chronic
Keywords: Hepatitis C, Chronic; Interferon-alpha; Hepatitis C Virus
MeSH Terms: conditions — Hepatitis C, Chronic; Hepatitis C | interventions — peginterferon alfa-2a

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- PEGASYS 180 µg Q1W + ribavirin* for 48 weeks (Active Comparator): Pegasys 180 µg Q1W(subcutaneous injection)+Ribavirin, multiple doses(48)
  Interventions: Biological: PEGASYS 180 µg Q1W
- P1101 180 µg Q1W + ribavirin* for 48 weeks (Experimental): P1101 180 µg Q1W(subcutaneous injection)with Ribavirin, multiple doses
  Interventions: Biological: P1101 180 µg Q1W, 48 doses
- P1101 270 µg Q1W + ribavirin* for 48 weeks (Experimental): P1101 270 µg Q1W(subcutaneous injection)+Ribavirin, multiple doses
  Interventions: Biological: P1101 270µg Q1W, 48 doses
- P1101 450 µg Q2W + ribavirin* for 48 weeks (Experimental): P1101 450 µg Q2W(subcutaneous injection)+Ribavirin, multiple doses
  Interventions: Biological: P1101 450µg Q2W, 24 doses

INTERVENTIONS:
Biological: PEGASYS 180 µg Q1W — 48 doses, solution, 48 weeks
  Arms: PEGASYS 180 µg Q1W + ribavirin* for 48 weeks
Biological: P1101 180 µg Q1W, 48 doses — 48 doses, solution, 48 weeks
  Arms: P1101 180 µg Q1W + ribavirin* for 48 weeks
Biological: P1101 270µg Q1W, 48 doses — 48 doses, solution, 48 weeks
  Arms: P1101 270 µg Q1W + ribavirin* for 48 weeks
Biological: P1101 450µg Q2W, 24 doses — 24 doses, solution, 48 weeks
  Arms: P1101 450 µg Q2W + ribavirin* for 48 weeks

SUMMARY:
Primary objectives:

The purpose of this study is to determine and compare the sustained virologic response (SVR, undetectable HCV RNA at Follow up week 24 (FW24)) across treatment groups.

To determine and compare the safety and tolerability of P1101 + Ribavirin across treatment groups.

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥18 years of age (≥ 20 years for subjects enrolled in Taiwan); subjects who are over 70 years of age must be in generally good health.
* Confirmed diagnosis of chronic hepatitis C (CHC) virus genotype 1 infection: (1) Positive for anti-HCV antibody or HCV RNA at least 6 months before screening, and positive for HCV RNA genotype 1 or anti-HCV antibody at the time of screening; or (2) Positive for anti-HCV antibody or HCV RNA genotype 1 at the time of screening with a liver biopsy consistent with chronic HCV infection (or a liver biopsy performed before enrollment with evidence of CHC disease, such as the presence of fibrosis).
* Compensated liver disease: with normal or elevated alanine aminotransaminase (ALT)/ aspartate aminotransferase (AST) (≤ 5 times the upper limit of normal), normal bilirubin level (< 2 mg/dL, except for Gilbert's syndrome), normal albumin, normal prothrombin time (PT) (INR< 1.3), no clinical symptoms or signs of cirrhosis or liver decompensation, and no evidence of cirrhosis as identified by ultrasound or any other procedures within 6 months before study entry.
* Treatment naïve: never received interferon, ribavirin or any other HCV treatment.
* No other form of chronic liver disease apart from chronic hepatitis C infection.
* Hemoglobin ≥ 13 g/dL in men or ≥ 12 g/dL in women, white blood cell (WBC) count ≥ 3,500/mm3, absolute neutrophil count (ANC) ≥ 1,500/mm3, platelet count ≥ 90,000/mm3; renal biochemistry estimated glomerular filtration rate (eGFR) > 60 mL/min.
* Be able to attend all scheduled visits and to comply with all study procedures.
* Be able to provide written informed consent.

Exclusion Criteria:

* Clinically significant illness or surgery within 4 weeks prior to dosing.
* Any clinically significant abnormality or abnormal laboratory test results found during medical screening besides serum ALT/AST (≤ 5 times the upper limit of normal).
* Any reason which, in the opinion of the investigator, would prevent the subject from participating in the study.
* Positive test for hepatitis B surface antigen (HBsAg) or human immunodeficiency virus (HIV) at screening.
* Clinically significant vital sign abnormalities at screening.
* Significant or major fundoscopic findings including but not limited to retinal exudates, hemorrhage, detachment, neovascularization, papilloedema, optic atrophy, microaneurysms and macular changes.
* History of significant alcohol or drug abuse within one year prior to the screening visit (alcohol consumption of more than fourteen units of alcohol per week [1 Unit = 150 mL of wine, 360 mL of beer, or 45 mL of 40% alcohol]) or refusal to abstain from alcohol or illicit drugs throughout the study.
* Pregnancy or, in women of child-bearing potential or in spouses of such women, unwillingness or inability to practice adequate contraception, defined as vasectomy in men, tubal ligation in women, or use of condoms and spermicides, or birth control pills, or intrauterine devices throughout the study.
* History of severe allergic or hypersensitivity reactions (like angioedema), specifically asthma, any known reaction to the study medication, allergic skin rash or other allergic reactions (like anaphylaxis), including severe drug allergies.
* Therapy with any systemic anti-viral, anti-neoplastic, and immunomodulatory treatment (including supraphysiologic doses of steroids and radiation) within 6 months prior to the first dose of study drug.
* Use of an investigational drug within the last 4 weeks from first dose of this study.
* Clinically significant gastrointestinal pathology (eg, chronic diarrhea, inflammatory bowel diseases), unresolved gastrointestinal symptoms (eg, diarrhea, vomiting), liver (other than CHC) or kidney disease (including but not limited to those with chronic renal failure on dialysis), or other conditions known to interfere with the absorption, distribution, metabolism, or excretion of the drug.
* Any clinically significant history or presence of major or poorly controlled psychiatric (including but not limited to those with severe depression, severe bipolar disorder, schizophrenia, suicidal ideation or history of suicidal attempt), neurological, cardiovascular, pulmonary (including but not limited to chronic obstructive lung disease), hematological, immunologic, endocrine, metabolic or other uncontrolled systemic disease, coagulation disorders or blood dyscrasias.
* A depot injection or an implant of any drug within 3 months prior to administration of study medication, other than contraception.
* Donation of plasma (500 mL) within 7 days prior to drug administration. Donation or loss of whole blood (excluding the volume of blood that will be drawn during the screening procedures of this study) prior to administration of the study medication as follows: 50 mL to 499 mL of whole blood within 30 days, or more than 499 mL of whole blood within 56 days prior to drug administration.
* Body organ transplant and are taking immunosuppressants.
* History of malignant disease, including solid tumors and hematologic malignancies (except basal cell and squamous cell carcinomas of the skin that have been completely excised and are considered cured); however, subjects who are cancer survivors not on maintenance therapy had no malignant diseases history within the past 5 years could be recruited.
* History of opportunistic infection (eg, invasive candidiasis or pneumocystis pneumonia).
* Serious local infection (eg, cellulitis, abscess) or systemic infection (eg, septicemia) within the 3 months prior to screening.
* Inability to comprehend the written consent form.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2011-10-18 (Actual); Primary Completion 2016-11-22 (Actual); Study Completion 2016-11-22 (Actual)

PRIMARY OUTCOMES:
Sustained Virologic Response | Follow up week 24 across treatment groups
  Percentage of subjects with sustained virologic response (SVR, undetectable HCV RNA at follow up week 24) across treatment groups.

CONTACTS AND LOCATIONS:
Overall Officials: Kuan-Chiao Tseng, MD, Sc.D., Study Director — PharmaEssentia Corp.
Locations (13):
- Taiwan (13):
  - Changhua Christian Hospital, Changhua
  - National Taiwan University Hospital - Yunlin, Douliu
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - Chang Gung Medical Foundation - Kaohsiung, Kaohsiung City
  - Chang Gung Medical Foundation - Keelung, Keelung
  - Chang Gung Medical Foundation - Linkou, Linkou District
  - Far Eastern Memorial Hospital, New Taipei City
  - Buddhist Tzu Chi General Hospital, Sindian City
  - China Medical University Hospital, Taichung
  - Taichung Veterans General Hospital, Taichung
  - National Taiwan University Hospital, Taipei
  - Cathay General Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei

REFERENCES:
- [Result] Lin HH, Hsu SJ, Lu SN, Chuang WL, Hsu CW, Chien RN, Yang SS, Su WW, Wu JC, Lee TH, Peng CY, Tseng KC, Qin A, Huang YW, Chen PJ. Ropeginterferon alfa-2b in patients with genotype 1 chronic hepatitis C: Pharmacokinetics, safety, and preliminary efficacy. JGH Open. 2021 Jul 10;5(8):929-940. doi: 10.1002/jgh3.12613. eCollection 2021 Aug. PMID 34386602
- See also: Related Info — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC8341194/